CLINICAL TRIAL: NCT01758406
Title: Therapeutic Outcome of Intracoronary Transplantation of Autologous Cardiac Stem Cells in Patients With Ischemic Heart Failure: Randomized Double Blind Clinical Trial
Brief Title: Transplantation of Autologous Cardiac Stem Cells in Ischemic Heart Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Heart-003
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: Cardiac stem ce heart failure cardiac function intracoronary transplantation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cardiac stem cell transplantation (Experimental): The patients with heart failure that underwent cardiac stem cell transplantation.
  Interventions: Biological: Intracoronary injection
- Placebo (Placebo Comparator): The patients with heart failure that underwent placebo injection.
  Interventions: Biological: Intracoronary injection of Placebo

INTERVENTIONS:
Biological: Intracoronary injection — stem cell transplantation
  Other Names: autologous cardiac stem cell intracoronary injection
  Arms: cardiac stem cell transplantation
Biological: Intracoronary injection of Placebo — Injection of Placebo via coronary arteries in patients with heart failure.
  Arms: Placebo

SUMMARY:
This study is a prospective, randomized, double blind , controlled trial to assess the efficacy of intracoronary transplantation of autologous cardiac stem cells in 50 patients with ischemic heart failure.

DETAILED DESCRIPTION:
Heart failure is a common, costly, disabling, and potentially deadly condition. Heart transplantation is the ultimate approach to treating heart failure, but this is costly and excludes patients who are poor candidates for transplantation given their co morbidities, or for whom a donor organ is unavailable. Currently, there is no effective intervention to regenerate dead heart muscle after a heart attack. Our hypothesis is that CSCs regenerates myocardium. In this study all eligible patients are randomly allocated into two study groups by a permuted block randomization method: group A (case group) received 5-10 millions autologous cardiac stem cells, group B (control group) just received placebo. They follow up for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 1- EF≤40 (by Echocardiography) 2- Not responding to standard therapies for heart failure >1m 3- NYHA class ≥ III 4- Myocardial infarction due to coronary artery atherosclerotic disease 5-An area of regional dysfunction, i.e., hypokinetic, akinetic, or dyskinetic (echocardiography or MRI) 6-No HIV/Viral hepatitis 7-Normal liver function (SGPT < 3 times the upper reference range) 8-No or controlled diabetes (hemoglobin A1C < 8.5%) 9- Ability to provide informed consent and follow-up with protocol procedures

Exclusion Criteria:

* 1 prior ICD placement(<2w)/Sustained ventricular arrhythmias 2-Cardiogenic shock 3- pregnancy and Child-bearing 4- Congenital / valvular heart disease

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
death | 18months
  evaluation the rate of patients mortality after cardiac stem cell transplantation.
arrhythmia | 18months
  Evaluation rate of arrhythmia after cardiac stem cell transplantation
hospitalization | 18 months
  Evaluation the rate of hospitalization after cardiac stem cell transplantation

SECONDARY OUTCOMES:
Ejectin fraction changes | 18months
  evaluation the elevation of ejection fraction in patients after cardiac stem cell transplantation.
Pro BNP changes | 18months
  Evaluation the reduction of Pro BNP in patients after cardiac stem cell transplantation.
NYHA functional class | 18months
  Evaluation the improvement of NYHA functional class in patients after cardiac stem cell transplantation.
6MW test | 18months
  Evaluation the improvement of 6MW test after cardiac stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan department of degenerative medicine; Ahmad Amin, MD, Study Director — Department of Heart failure,Shahid Rajaee Hospital; Farveh Vakilian, MD, Principal Investigator — Department of Heart failure , Imam reza hospital, Mashhad, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org